CLINICAL TRIAL: NCT05266300
Title: Implementation and Quality Assurance of DPYD-genotyping in Patients Treated With Fluoropyrimidines
Status: Completed | Type: Observational
Sponsor: University of Southern Denmark (Other)
Collaborators: Odense University Hospital (Other)
Responsible Party: Principal Investigator, Per Damkier, MD, ph.d. Clinical Professor,, University of Southern Denmark
Other Study IDs: R231-A14057
Record Dates: First submitted 2021-12-16; First posted 2022-03-04 (Actual); Last update posted 2022-11-01 (Actual); Status verified 2022-10

CONDITIONS: Adverse Drug Event; Colon Cancer; Breast Cancer; Pancreas Cancer; Rectal Cancer; Gastric Cancer; Oesophageal Cancer; Bile Duct Cancer
MeSH Terms: conditions — Drug-Related Side Effects and Adverse Reactions; Colonic Neoplasms; Breast Neoplasms; Pancreatic Neoplasms; Rectal Neoplasms; Stomach Neoplasms; Esophageal Neoplasms; Bile Duct Neoplasms | interventions — Dihydrouracil Dehydrogenase (NADP)

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Biospecimen Retention: Samples With DNA — Blood for phenotype analysis.(uracil and dihydrouracil concentrations)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Retrospective: Historic group. Patients treated in the historic control group did not receive DPYD-genotype before treatment with fluorouracil, capecitabine, tegafur. They received standard start doses of 5-FU, capecitabine, tegafur.
- Prospective: Participants enrolled in the prospective group will give a blood sample for immediate DPYD genotyping. Once the results from these tests are in, the treating oncologist have immediate access to the participant's genetic test results and can make dosing decisions/changes to the participant's chemotherapy prescription. The recommended starting doses for 5-FU, capecitabine, tegafur are.
  No DPYD-gene variant = normal starting dose (100%)
  1 DPYD-gene variant (heterozygous) = Reduced starting dose (50%) Homozygous for 1 DPYD variant or compound heterozygous (>1 variants) = Treatment with 5-FU, capecitabine, tegafur is not recommended .
  Interventions: Genetic: DPYD genotype

INTERVENTIONS:
Genetic: DPYD genotype — The SNPs included in this study are the following (dbSNP Reference SNP)
  rs3918290(c.1905+1G>A) rs67376798(c.2846A>T) rs55886062(c.1679T>G) rs56038477(75017182)/(c.1236G>A)
  Other Names: Dihydropyrimidine dehydrogenase (DPD) enzyme activity
  Groups: Prospective

SUMMARY:
The purpose of this study is to examine the benefits of a clinical implementation of a DPYD-genotype test to patients starting treatment with fluoropyrimidines (Fluorouracil (5-FU), capecitabine, tegafur).

DETAILED DESCRIPTION:
Patients with specific genetic mutations in the DPYD-gene have lower activity of the dihydropyrimidine dehydrogenase (DPD) enzyme, which is the rate-limiting enzyme in the metabolism of fluoropyrimidines. Fluoropyrimidines are commonly used as chemotherapeutic drugs and include 5-Fluorouracil, capecitabine, and tegafur. Patients with decreased DPD activity are at higher risk of serious adverse events when treated with standard doses of fluoropyrimidines

This study will examine the clinical implementation of the pre-emptive DPYD-genotype test. The test will analyze four of the most common genetic mutations(SNPs) in the DPYD-gene that leads to significant decreased DPD-activity

In patients with DPYD-variant mutations, the recommended starting dose is 50%. This dose reduction will possibly reduce the rate of serious adverse events. Patients who are homozygous or compound heterozygous for a DPYD-mutation will not be treated with fluoropyrimidines due to the high risk of fatal adverse effects.

Aim To reduce the overall incidence of severe adverse reactions(grade >= 3) to chemotherapy regimens containing 5-FU, capecitabine, or S1 in an unselected population of colorectal, non-colorectal GI cancer, or breast cancer patients through pre-emptive DPYD-genotyping.

Design The investigators will conduct an open clinical trial using historical controls. The investigators will implement pre-emptive genotype testing of about 1000 consecutive patients subject to 5-FU, capecitabine, or S1 treatment for colorectal, non-colorectal GI, or breast cancer. The investigators will use a historical control group of about 500 consecutive similar patients.

Genotype and Phenotype Patients included in the study who are genotyped for DPYD will have blood collected for a post hoc phenotype test. The blood samples will be used to measure levels of uracil.

Some patients in the historic cohort have donated blood to an independent biobank at the time of their cancer treatment. These samples will be used for post hoc DPYD-genotype analysis after the necessary ethical approvals.

Cost-effectiveness An economic analysis will be undertaken to examine if implementing the DPYD-genotype is cost-effective.

ELIGIBILITY:
Inclusion Criteria:

* Patients with cancer that are eligible for systemic treatment with 5-FU, capecitabine, or tegafur.

Exclusion Criteria:

* Patients that earlier have been treated with 5-FU, capecitabine, or tegafur

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Cancer patients treated at The Department of Oncology at Odense University Hospital (OUH)
Sampling Method: Non-Probability Sample
Enrollment: 722 (Actual)
Dates: Start 2020-09-01 (Actual); Primary Completion 2022-06-01 (Actual); Study Completion 2022-10-01 (Actual)

PRIMARY OUTCOMES:
Adverse events | Up to 6 months
  Rate of grade 3-5 adverse events (CTCAE) Version 5.0

SECONDARY OUTCOMES:
5-FU or capecitabine or S1-related mortality, all patients | Up to 6 months
  Rate of mortality related to adverse drug reaction
5-FU or capecitabine or S1-related mortality, DPYD variant carriers | Up to 6 months
  Rate of mortality related to adverse drug reactions in patients with a DPYD gene variant.
Overall mortality, all patients | Up to 6 months
  Rate of mortality in all patients
Overall mortality, DPYD variant carriers | Up to 6 months
  Rate of mortality in patients with DPYD-variants.
Length of hospital stay | Up to 6 months
  Number of days participants is admitted to the hospital.
Rate of discontinuation of fluoropyrimidines due to adverse events | Up to 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Per Damkier, MD, PhD, Principal Investigator — University of Southern Denmark
Locations (1):
- The Department of Oncology at University of southern denmark, Odense, Region Syddanmark, Denmark

IPD SHARING:
Plan to Share IPD: No